CLINICAL TRIAL: NCT04129060
Title: Health of the Cholinergic System and Risk for Alzheimer's Disease in Postmenopausal Women
Brief Title: Cholinergic Health After Menopause (CHAMP)
Acronym: CHAMP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Julie Dumas, Associate Professor, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00000581
Record Dates: First submitted 2019-10-09; First posted 2019-10-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Postmenopausal Symptoms; Aging; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Cholinergic Antagonists

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo-controlled trial of the effects of nicotinic blockade on working memory performance and brain activation in healthy postmenopausal women.
Who Masked: Participant, Investigator
Masking Description: Medication will be administered double blind. The investigators, nurses working on the project, and participants will not know which drug they receive on any study day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mecamylamine Challenge (Experimental): One of the two study days will be the oral mecamylamine.
  Interventions: Drug: Cholinergic antagonist
- Placebo Challenge (Experimental): One of the two study days will be the oral placebo.
  Interventions: Drug: Cholinergic antagonist

INTERVENTIONS:
Drug: Cholinergic antagonist — The cholinergic antagonist drug mecamylamine will be administered as a a 20 mg oral pill and matching placebo

SUMMARY:
Women are at increased risk for Alzheimer's disease (AD). Notably at menopause, some women experience a change in cognition. However, not all women experience negative effects of menopause on cognition. The cognitive changes that occur at menopause have not yet been connected to late life risk for pathological aging including AD. Thus, understanding the neurobiological factors related to individual differences in cognition at menopause is critical for understanding normal cognitive aging and for determining risk for pathological aging. The challenge in understanding the role of estrogen loss on the risk for AD is the long lag time between the hormonal changes at menopause and the clinical manifestations of AD. Thus, identifying how the hormone changes after menopause are related to AD risk will alter the risk calculus for postmenopausal women in the future.

The novel study proposed here will examine an established AD-related neurotransmitter-based mechanism that may also underlie cognitive changes after menopause. The investigators propose that the change in the hormonal milieu at menopause interacts with the cholinergic system and other brain pathologies to influence a woman's risk for cognitive decline. Preclinical studies have shown that estrogen is necessary for normal cholinergic functioning and its withdrawal leads to cholinergic dysfunction and cognitive impairment. It is important to determine whether menopause-related cognitive changes correlate with both cholinergic functional integrity and established AD biomarkers that portend increased risk for late-life cognitive impairment or dementia. This study will examine brain functioning following cholinergic blockade to separate individuals into those who are able to compensate for the hormone change after menopause and those who are not. The investigators hypothesize women with poor compensation have increased sensitivity to cholinergic blockade by showing poor performance on a cognitive task, altered brain activation, and decreased basal forebrain cholinergic system (BFCS) volume. These cholinergic markers will be related to menopausal factors associated with poor cognition and biomarkers of AD.

Specific Aim 1 is to examine cholinergic functional "integrity" by measuring working memory performance, functional brain activation, and BFCS structure in postmenopausal women. Specific Aim 2 will examine whether individual differences in menopause-relevant symptoms and known AD biomarkers are related to cognition and brain activation after anticholinergic challenge.

The public health significance of this study is that it will identify individual difference factors that are associated with cognitive performance changes after menopause and their relationship to structural, functional, and biomarker evidence of risk for later life cognitive dysfunction. Knowledge of these factors will serve to advance personalized future risk-mitigation strategies for women including hormonal, medication, cognitive remediation, etc. that will be the subject of further research.

DETAILED DESCRIPTION:
The brain is a major target for circulating gonadal steroids and the change in hormone levels after menopause is likely to have implications for cognitive functioning. A number of clinical and preclinical studies have linked gonadal steroids and cognition (e.g.1,2) and it has been hypothesized that menopause has detrimental effects on cognition that are over and above the expected effects of normal aging. While menopause results in reproductive senescence, most of the symptoms of menopause are neurological3. However, evidence for changes in brain functioning after menopause is equivocal. Some studies found that cognitive performance after menopause decreased in domains such as memory, attention, problem solving, and motor skills from pre-menopausal levels (e.g.1,4,5). As many as 60% of women reported undesirable memory changes at mid-life6. Other studies have not found changes in cognition after menopause (e.g.7-9) and not all women experience negative effects of menopause on cognition10. However, women have a higher risk of dementia compared to men11 and many hypotheses identify the sex differences in gonadal steroids and the hormone change at menopause as related to risk for Alzheimer's disease (AD) and/or dementia. The challenge in understanding the role of estrogen loss on the risk for AD is the long lag time between the hormonal changes at menopause and the clinical manifestations of AD. Thus, identifying how the hormone changes after menopause are related to AD risk will alter the risk calculus for postmenopausal women in the future. In addition, the neurobiological processes underlying how the change in the hormonal environment at menopause influences brain functioning, what factors are responsible for individual differences in cognition after menopause, and what menopause-related symptoms are associated with risk for dementia are not well understood.

One mechanism hypothesized to be responsible for cognitive changes post menopause is the effect of decreased estradiol on the functioning of neurotransmitter systems that support cognition. The importance of the estrogen-cholinergic system interaction for cognition has been demonstrated across a number of model systems from rats12 to non-human primates13 to humans14. The investigators have shown that estrogen's interaction with the cholinergic system is important for cognitive functioning in postmenopausal women14-16. What has not not yet shown is how change in cholinergic system functioning as a result of menopause is related to menopausal signs/symptoms that influence cognition as well as AD biomarkers like amyloid, tau, and neurodegeneration. These are important relationships to understand and may lead to individual risk profiles that can be observed earlier in the aging process while treatment and prevention strategies may be effective.

This project will investigate the role of cholinergic system in cognitive functioning in women after menopause. We have been examining the interaction of the neurotransmitter acetylcholine with hormones after menopause for a number of years14-16. In these studies with intensive repeated measures designs where the sample sizes were relatively small, findings generally showed no benefit of estrogen therapy alone for cognition in normal women post menopause. However, if the investigators induced a temporary impairment in the cholinergic system, the beneficial effect of estradiol became manifest15 and this was more prominent in younger postmenopausal women aged 50-60 compared to older women aged 70-8014. Furthermore, these studies showed significant heterogeneity of individual responses with roughly 50% of women showing either compensatory or impaired responses suggesting individual differences in risk profile (see preliminary data). What has not yet demonstrated is how the sensitivity of the cholinergic system to temporary blockade is related to menopause symptoms and known AD biomarkers that are associated with increased risk for AD development or frank dementia.

The investigators propose that cholinergic antagonist drugs can be used to expose the effects of menopause on cognitive functioning. Decreased cognitive performance during a temporary cholinergic blockade "lesion" may be an indicator of susceptibility to the negative effects of hormone withdrawal on the brain and risk for age-related cognitive impairment and/or dementia. The study proposed here will be the first to link cholinergic sensitivity to biomarkers of neurodegeneration and AD pathology. Specifically, the study will investigate working memory performance and brain activation during a cholinergic antagonist challenge compared to placebo and examine how factors associated with menopause like gonadal steroids, autonomic symptoms, mood, and sleep as well as known biomarkers associated with Alzheimer's disease (e.g. age, subjective cognitive complaints, hippocampal and basal forebrain volume, beta amyloid, and tau load) combine to predict which women are likely to experience cognitive impairment during the cholinergic challenge procedure.

The results from this study will further the understanding of the neurotransmitter-based mechanisms responsible for cognitive changes after menopause and how these may predict late life cognitive dysfunction. After an examination of the neurobiology underlying the cognitive change at menopause, future studies can develop strategies to mitigate pathological processes that are enhanced by the menopausal hormone change.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-70 years
* Postmenopausal
* Nonsmokers
* Not taking hormone therapy, selective serotonin uptake inhibitors (SSRIs(, phytoestrogens, selective estrogen receptor modulators (SERMS), or antiestrogen medications and will be at least one year without such treatment
* Physically healthy
* No cardiovascular disease other than mild hypertension. Subjects will also not have current untreated or unremitted Axis I or II psychiatric or cognitive disorders (see screening below).
* Intelligence quotient (IQ) in the normal range >80
* Normal neuropsychological test performance

Exclusion Criteria:

* Mild Cognitive Impairment (MCI) or dementia - Montreal Cognitive Assessment <26, Mattis Dementia Rating Scale <130, and Global Deterioration Scale >2
* History of cancer treatment with cytotoxic and/or ongoing (current) maintenance targeted chemotherapy
* Blood pressure > 160/100 (untreated)
* Untreated thyroid disease
* Significant cardiovascular disease
* Asthma or chronic obstructive pulmonary disease (COPD)
* Active peptic ulcer
* Hyperthyroidism
* Epilepsy
* Current untreated or unremitted Axis I psychiatric disorders
* Use of medications that are on our prohibited medications list

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Dependent (BOLD) functional magnetic resonance imaging (fMRI) | Two hours post drug administration
  BOLD fMRI signal will be measured while each participant performs the N-back test.
Working Memory Performance | Two hours post drug administration
  We will assess performance on the N-back test of working memory test.
Basal Forebrain Cholinergic System Volume | Two hours post drug administration
  We will measure basal forebrain cholinergic system volume from the T1 images acquired during the MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Dumas, Ph.D., Principal Investigator — University of Vermont; Paul A Newhouse, M.D., Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
We will make data available at the end of the study after the blind has been broken. We will use a federally available database like the National Institutes of Mental Health (NIMH) Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available at the end of the study
Access Criteria: We will have the same requirements for data sharing as the NDA has run by the NIMH.